CLINICAL TRIAL: NCT07195344
Title: Influence of Patient's Morphological Characteristics on Pharmacokinetic and Toxicity of Trastuzumab-Deruxtecan Administered for Metastatic Breast Cancers
Brief Title: Study Aiming to Compare the Plasma Exposure of the Payload (Free-DXd) in Patients Treated by T-DXd for Locally Advanced or Metastatic Breast Cancer According to Their BMI.
Acronym: TDXdose
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25SEIN06
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced or Metastatic Breast Cancers
Keywords: Locally or metastatic Breast Cancer; HER2 low-expressed; HER2 over-expressed/amplified; Trastuzumab-Deruxtecan; Body Mass Index; Pharmacokinetics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with locally advanced or metastatic breast cancer starting T-DXd as standard treatment (Other)
  Interventions: Biological: Pharmacokinetics blood samples

INTERVENTIONS:
Biological: Pharmacokinetics blood samples — Blood samples will be collected at different time points during the first four treatment cycles and at the end of T-DXd treatment or at 24 months after inclusion in case of T-DXd continuation beyond this time period.

SUMMARY:
This is a multicenter, prospective, non-randomized, open-label, pharmacokinetic study, aiming to compare the plasma exposure of the payload (free-DXd) in patients treated by T-DXd for locally advanced or metastatic breast cancer according to their BMI.

The primary objective is to compare plasma exposition of the payload (free-DXd) between overweight or obese (BMI>25) and normal weight (BMI≤25) breast cancer patients during the first 3 cycles of Trastuzumab-Deruxtecan (T-DXd).

A total of 210 patients will have to be enrolled in this study with the following repartition:

N = 105 patients with a BMI ≤ 25 (normal weight patients). N = 105 patients with a BMI > 25 (overweight or obese patients) with at least 30 obese patients (BMI>30).

ELIGIBILITY:
Inclusion Criteria:

1. Women (or men) aged ≥ 18 years on the day of signing the informed consent with histologically proven breast cancer.
2. Metastatic or locally advanced breast cancer with overexpression/amplification HER2 (IHC +++ or ++ and positive-hybridation in situ) or low HER2 expression (IHC + or ++ and negative-hybridation in situ) and may be ultra-low (in first line, in case of approval).
3. Patient eligible for Trastuzumab-Deruxtecan (T-DXd).
4. Concomitant administration of pertuzumab may be accepted in case of approval in first line for HER2- overexpressed/amplified locally advanced or metastatic breast cancer.
5. Female subjects of childbearing potential must have a negative pregnancy test within 72 hours prior to receiving the first dose of study treatment.
6. Female subjects of childbearing potential must be willing to follow at least one method of contraception or be surgically sterile, or abstain from heterosexual activity for the duration of the study and until 7 months after the last dose of study treatment. Subjects of childbearing potential are those who have not been surgically sterilized and who had menstruation in the last 12 months.

   Note: Abstinence is acceptable if it is the subject's usual lifestyle and preferred method of contraception.
7. Male subjects must agree to use at least one method of contraception for the duration of the study and until 4 months after the last dose of study treatment.

   Note: Abstinence is acceptable if it is the subject's usual lifestyle and preferred method of contraception.
8. Signed written informed consent.
9. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol.
10. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Peripheral venous access making blood samples difficult.
2. Patients unable to receive T-DXd treatment at a dose of 5.4 mg/kg in cycle 1 (whatever the reason)
3. Patients with known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
4. Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the study.
5. Patient pregnant, or breast-feeding.
6. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
7. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).
8. Concurrent participation in an experimental drug study.
9. Patient with a known history of hypersensitivity to the active substance of T-DXd or to any of the excipients listed in the SmPC of T-DXd.
10. Patient with severe hepatic impairment defined by TGO and/or TGP > 5 x ULN and Total bilirubin > 1.5 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | From the 1st cycle of T-DXd (C1D1) to the end of the 3rd cycle of T-DXD (each cycle is 21 days) treatment or until an event (interruption or dose concession for toxicity) if it occurs before the 3rd cycle.
  Plasma exposure of free-DXd (payload) will be measured by the cumulative AUC (Area under the concentration vs. time curve) over the first 3 cycles or until an event (interruption or dose concession for toxicity) divided by the number of corresponding cycles.
  These AUCs will be determined by Bayesian estimation (Posthoc values) using a non-linear mixed-effects approach.

SECONDARY OUTCOMES:
Safety: toxicities will be assessed using the NCI-CTCAE Version 5.0. | From enrollment to the end of patient participation up to 24 months after inclusion
Efficacy: Progression Free Survival (PFS) | From inclusion until progression or death up to 24 months after inclusion
  Progression Free Survival (PFS) is defined as the time from inclusion until progression or death; patients alive and without documented progression at last follow-up news are censored at this date or at initiation of new anticancer treatment (if applicable).
Secondary pharmacokinetic criteria | From C1D1 to definitive stop of T-DXd treatment up to 24 months after inclusion
  A population PK model will be performed to quantify the impact of several patient characteristics: morphological data (weight, height, BMI, lean mass, etc.), biological data (inflammation markers, albuminemia, liver enzymes, etc.), demographic data (age), on the PK parameters (elimination clearance, volume of distribution) of T-DXd and free-DXd.
Body composition parameters | From enrollment to tumor assessment before C9D1 at 6 months of T-DXd treatment (each cycle is 21 days).
  Skeletal muscle mass index or density and lean body mass before treatment initiation and during the active treatment phase (at 3 months tumor assessment before C5D1 and at 6 months; tumor assessment before C9D1) using the "Cassandra" algorithm.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Institut de Cancérologie de l'Ouest - Site Angers, Angers
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU de Nîmes, Nîmes
  - Institut Curie - Site Paris, Paris
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest - Site Saint Herblain, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - IUCT-O, Toulouse